CLINICAL TRIAL: NCT06701162
Title: TRANSVERSE ABDOMINAL PLANE BLOCK VS. ILIO-INGUINAL ILIO-HYPOGASTRIC BLOCK in PEDIATRIC INGUINAL SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Head of the Department of Anesthesiology and Critical Care, Tunis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 012020
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Analgesia; Ultrasound Guided Block
Keywords: Transverse abdominal plane bloc; pain; analgesia; ultrasound; children
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: The patients were randomly assigned into two groups to receive after a standardized induction of general anesthesia either an ultrasound-guided TAP block or IIIH block with bupivacaine 0.3 ml/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP group (Other): Uktrasound-guided TAP block
  Interventions: Procedure: Ultrasoud-guided TAP block
- IIIH block (Other): Ultrasound-guided Ilio-inguinal Ilio-Hypogastric Block
  Interventions: Procedure: Ultrasound-guided Ilio-inguinal Ilio-Hypogatric block

INTERVENTIONS:
Procedure: Ultrasoud-guided TAP block — the ultrasound probe was placed at the mid-axillary line, and the needle was inserted into the space between the internal oblique and transverse muscles, splitting the inter-muscular fascia after injection of local anesthetic.
  Arms: TAP group
Procedure: Ultrasound-guided Ilio-inguinal Ilio-Hypogatric block — the ultrasound probe was positioned transversely on the abdominal wall at the contact point of the anterosuperior iliac spine. The needle was inserted into the space between the internal oblique and transverse muscles, causing separation of the intermuscular fascia layers upon injection of the anesthetic mixture
  Arms: IIIH block

SUMMARY:
The ilio-inguinal ilio-hypogastric (IIIH) nerve block remains the gold standard analgesic technique after inguinal surgery in children. Transverse abdominal plane (TAP) block has been reported to provide effective analgesia after lower abdominal surgery in adults. The aim of our study was to compare the analgesic effect of ultrasound-guided TAP block to IIIH nerve block after inguinal surgery in children.

DETAILED DESCRIPTION:
The study aimed to compare the analgesic effect of ultrasound-guided transverse abdominal plane (TAP) block to ilio-inguinal ilio-hypogastric (IIIH) nerve block in children after inguinal surgery. This prospective, randomized study included children aged six months to twelve years, classified as ASA I or II, scheduled for elective unilateral inguinal surgery. Participants received either a TAP block or an IIIH block with bupivacaine following standardized induction of general anesthesia. Analgesics were not systematically administered post-induction. Postoperative pain was monitored for six hours in the hospital, and if the CHEOPS score exceeded 7, paracetamol was administered, with nalbuphine as a secondary option if needed. At home, parents assessed pain using the PPMP score, administering paracetamol and ibuprofen if necessary. Primary outcomes included postoperative analgesia quality, determined by time to first analgesic requirement and the need for analgesics at hospital and home. Secondary outcomes measured included block performance duration, parental satisfaction, and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 12 years
* ASA physical status 1 or 2
* Scheduled for unilateral inguinal surgery

Exclusion Criteria:

* Children scheduled for bilateral surgery or associated procedures (e.g., circumcision)
* Parental refusal

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Quality of postoperative analgesia : PPMP score | 24 h after surgery
  The quality of postoperative analgesia described by the pain score : Postoperative Pain Measure for Parents (PPMP) score, minimum value is 0 , maximum value 10 , a value higher than 6 indicates a major pain .

SECONDARY OUTCOMES:
Block execution time | From the beginning of the practice of the block to the end
Complications related to the techniques of nerve block | Perioperative
  Complications related to local anesthetics or block technique such as hematoma, spread of local anesthetic to the femoral nerve, intraperitoneal injection ...

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza hospital, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided